CLINICAL TRIAL: NCT07284121
Title: A Non-Interventional, Multicenter, Multicohort Study to Evaluate Patient-Reported Satisfaction, Effectiveness, and Safety of Subcutaneous Atezolizumab in Participants Treated in Routine Clinical Practice
Brief Title: A Study to Evaluate Patient-Reported Satisfaction, Effectiveness, and Safety of Atezolizumab in Participants Treated in Routine Clinical Practice
Status: Recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MO45893
Record Dates: First submitted 2025-11-21; First posted 2025-12-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer, Hepatocellular Carcinoma
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Hepatocellular | interventions — atezolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Early Non-small Cell Lung Cancer (NSCLC): Participants diagnosed with early-stage NSCLC following complete resection and platinum-based chemotherapy with Programmed Cell-Death Ligand 1 (PD-L1) expression of >= 50% on Tumor Cell (TC).
  Interventions: Drug: Atezolizumab
- Cohort 2: Metastatic NSCLC: Participants diagnosed with metastatic NSCLC with PD-L1 expression of >= 50% on TC who have not received prior systemic therapy for metastatic disease.
  Interventions: Drug: Atezolizumab
- Cohort 3: Extensive stage small cell lung cancer (ES-SCLC): Participants diagnosed with ES-SCLC who have not previously been treated.
  Interventions: Drug: Atezolizumab
- Cohort 4: Hepatocellular Carcinoma (HCC): Participants diagnosed with advanced or unresectable HCC who have not received prior systemic therapy.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at the discretion of the treating physician and independently of participation in this study.
  Other Names: Tecentriq

SUMMARY:
This is a non-interventional, multi-country, multi-centre, multicohort, primary data collection study, designed to assess patients' reported satisfaction with Atezolizumab Subcutenous (SC) treatment and Health-related Quality of Life (HRQoL), as well as the effectiveness and safety of Atezolizumab SC in participants treated for selected approved indications in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have one of the following confirmed diagnoses for which atezolizumab is approved in the local SmPC:

  * Early stage NSCLC following complete resection and platinum-based chemotherapy with a high risk of recurrence and PD-L1 expression on ≥ 50% of TC and with no EGFR-mutant or ALK-positive NSCLC
  * Metastatic stage NSCLC with PD-L1 expression on ≥ 50% TC or ≥ 10% tumor infiltrating immune cells (IC) and with no EGFR-mutant or ALK-positive NSCLC not previously treated
  * Extensive-stage small cell lung cancer (ES-SCLC) not previously treated
  * Advanced or unresectable HCC not previously treated with systemic therapy
* Should not have received > 4 prior cycles of IV Atezolizumab

Exclusion Criteria:

* Not receiving treatment with Atezolizumab according to standard of care and in line with the current SmPC or local labelling
* Receiving concomitant systemic anticancer therapy at the time of initiation of Atezolizumab or an Atezolizumab-containing regimen for treatment of the same disease, as per label
* Receiving treatment with Atezolizumab as part of a clinical trial, pre-approval access program, compassionate use program, expanded use program, post-trial access program, or continued access program
* Unwilling to complete questionnaires related to treatment satisfaction and treatment-related quality of life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with early-stage NSCLC following complete resection and platinum-based chemotherapy with PD-L1 expression of >= 50% on TC, participants diagnosed with metastatic NSCLC with PD-L1 expression of ≥ 50% on TC who have not received prior systemic therapy for metastatic disease, participants diagnosed with ES-SCLC who have not previously been treated, and participants diagnosed with advanced or unresectable HCC who have not received prior systemic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Therapy Administration Satisfaction Questionnaire Subcutaneous (TASQ-SC) Score | At Cycle 2 and Cycle 3 (each cycle duration/length is 3 weeks)

SECONDARY OUTCOMES:
Overall Survival (OS) | Index date up to approximately 3.5 years
OS at 2 Years | After Index date up to 2 years
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) Score | Baseline or Index date
Percentage of Participants With Adverse Events | Up to approximately 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (80):
- Austria (4):
  - Landesklinikum Krems, Krems
  - Ordensklinikum Linz Elisabethinen, Linz
  - Krankenhaus Nord - Klinik Floridsdorf, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (2):
  - CHU HELORA - Hôpital de la Louvière - Site Jolimont, Haine-Saint-Paul
  - CHU UCL Mont-Godinne, Mont-godinne
- Bulgaria (6):
  - Multiprofile Hospital for Active Treatment Uni Hospital, Panagyurishte
  - Complex Oncological Center-Ruse EOOD, Rousse
  - Tokuda Hospital, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - MBAL Serdika EOOD, Sofia
  - MHAT SofiaMed, Sofia
- Italy (22):
  - Presidio Ospedaliero Vito Fazzi, Lecce, Apulia
  - AORN Ospedali dei Colli Ospedale Monaldi, Napoli, Campania
  - Az. Osp. Cardarelli, Napoli, Campania
  - A.O. Universitaria Policlinico Di Modena, Modena, Emilia-Romagna
  - Ospedale Provinciale Santa Maria Delle Croci, Ravenna, Emilia-Romagna
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Università Campus Bio-Medico di Roma, Rome, Lazio
  - IRCCS AOU San Martino - IST, Genoa, Liguria
  - Humanitas Gavazzeni, Bergamo, Lombardy
  - Fondazione IRCCS Ospedale Maggiore Policlinico, Milan, Lombardy
  - Ospedale Maggiore Policlinico, Milan, Lombardy
  - Asst Santi Paolo E Carlo, Milan, Lombardy
  - Ente Ecclesiastico Ospedale Generale Regionale F Miulli, Acquaviva Delle Fonti, Piedmont
  - A.O.U. Maggiore della Carità, Novara, Piedmont
  - Azienda Ospedaliero Universitaria Di Sassari, Sassari, Sardinia
  - Humanitas Istituto Clinico Catanese S.p.A, Misterbianco (CT), Sicily
  - A.O.U. Policlinico Paolo Giaccone, Palermo, Sicily
  - Casa di Cura La Maddalena, Palermo, Sicily
  - Azienda Sanitaria Territoriale Pesaro Urbino (AST PU) - Ospedale Santa Croce;UOC Oncologia - Stabilimento di Fano, Fano (PU), The Marches
  - Ospedale Santa Chiara, Trento, Trentino-Alto Adige
  - Ospedale dell'Angelo, Mestre, Veneto
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona, Veneto
- Poland (6):
  - Narodowy Instytut Onkologii - Panstwowy Instytut Badawczy, Oddzia? w Krakowie, Krakow
  - Uniwersytecki Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Warminsko-Mazurskie Centrum Chorób P?uc w Olsztynie, Olsztyn
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii w Poznaniu, Poznan
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka, Słupsk
  - NU-MED Centrum Diagnostyki i Terapii Onkologicznej, Tomaszów Mazowiecki
- Romania (7):
  - Institutul Clinic Fundeni Bucuresti, Bucharest
  - Institutul Regional de Gastroenterologie si Hepatologie Prof. Dr. Octavian Fodor, Cluj-Napoca
  - Spitalul Clinic Jude?ean de Urgen?? Sfântul Apostol Andrei Galati;oncology, Galati
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Municipal Ploiesti, Ploieşti
  - Spitalul Judetean de Urgenta Satu Mare, Satu Mare
  - Oncomed SRL, Timișoara
- Spain (30):
  - Complejo Hospitalario Torrecardenas, Almería, Almeria
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Sant Joan de Deu de Manresa;Servicio oncologia, Manresa, Barcelona
  - Hospital Universitario Puerto Real, Puerto Real, Cadiz
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, LA Coruna
  - Hospital Clínico Universitario Valladolid;servicio de digestivo, Valladolid, Madrid
  - Hospital Univ. Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Complejo Hospitalario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Tenerife
  - Hospital de Cruces, Bilbao, Vizcaya
  - Hospital Universitario de Cruces;servicio de digestivo, Vizcaya, Vizcaya
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General de Alicante;servicio de digestivo, Alicante
  - Hospital General Univ. de Alicante, Alicante
  - Hospital de Badajoz, Badajoz
  - Hospital Clinic I Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital Universitario San Cecilio, Granada
  - Hospital General Universitario de Guadalajara, Guadalajara
  - Hospital General Universitario J.M Morales Meseguer, Murcia
  - Hospital Virgen de Arrixaca;servicio de digestivo, Murcia
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Virgen del Rocio;Servicio de digestivo, Seville
  - Hospital de Toledo;Servicio de digestivo, Toledo
  - Hospital de Toledo;servicio de oncologia, Toledo
  - Hospital Arnau de Vilanova (Valencia) Servicio de Oncologia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - James Cook University Hospital, Middlesbrough
  - James Paget University Hospitals NHS Foundation Trust, Norfolk

IPD SHARING:
Plan to Share IPD: No